CLINICAL TRIAL: NCT06893159
Title: REACHing Underserved and Undiagnosed Populations Living with Syphilis and HIV in Alberta, Saskatchewan, Manitoba and Northern Communities: "Test, Treat and Linkage to Culturally Appropriate Care"
Brief Title: Ayaangwaamiziwin Initiative: Carefulness and Preparedness
Acronym: AI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: REACH-SPOR-001
Record Dates: First submitted 2025-02-27; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-01

CONDITIONS: Point-of-Care Testing; HIV; Syphilis
Keywords: HIV; syphilis; Point-of-care; Point-of-care testing; POC testing; Community-based
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Intervention Model Description: Screening for HIV and syphilis infection using 3 point-of-care devices by healthcare providers and non-healthcare providers at community-based clinical sites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients (Experimental): Patients will be anyone presenting at the community site clinics for regular STI testing
  Interventions: Device: INSTI HIV-1/2 Antibody Test; Device: INSTI Multiplex HIV-1/2 Syphilis Antibody Test; Device: Multiplo Complete Syphilis (TP/nTP) Antibody Test
- Healthcare Professionals (No Intervention): Healthcare professionals (e.g., nurses) that will conduct patient intake, consent patients, provide POC testing (test operators), and provide treatment and linkage to care where necessary.
- Non-Healthcare Professionals (No Intervention): Non-Healthcare Professionals (e.g., health navigators that are peers with lived experiences) that will conduct community outreach, and for sites that are doing non-healthcare professional testing, the health navigators will conduct patient intake, consent patients, provide POC testing (test operators), and link patients to treatment where necessary.

INTERVENTIONS:
Device: INSTI HIV-1/2 Antibody Test — The INSTI HIV-1/HIV-2 Antibody Test is a single use, rapid, in vitro qualitative immunoassay for the detection of antibodies to Human Immunodeficiency Virus Type 1 and/or Type 2 (HIV-1/HIV-2) in human venipuncture whole blood, fingerstick blood, or plasma specimens. The test is intended for use by trained personnel in point of care and laboratory situations to aid in the diagnosis of HIV infections. If multiple rapid HIV tests are available, this test is suitable for use in appropriate multi-test algorithms.
  Arms: Patients
Device: INSTI Multiplex HIV-1/2 Syphilis Antibody Test — The INSTI MULTIPLEX HIV-1/2 Syphilis Ab Test is a single use, rapid, flow-through in vitro qualitative immunoassay for the detection of antibodies to Human Immunodeficiency Virus Type 1/ Type 2 and Treponema pallidum in human fingerstick blood and serum. The INSTI Multiplex Test is intended as an aid in the diagnosis of HIV1/2 and Syphilis infections in patients with signs and symptoms of HIV and Syphilis. The test is intended for use by trained personnel in medical facilities, clinical laboratories, emergency care situations, and physicians' offices as an in vitro diagnostic device capable of providing results in less than one minute. Although suitable for near-patient point-of-care (POC) testing, the INSTI Multiplex Test is not suitable for self-testing.
  Arms: Patients
Device: Multiplo Complete Syphilis (TP/nTP) Antibody Test — Multiplo Complete Syphilis (TP/nTP) Antibody Test (Multiplo® TP/nTP) is a single use, manually performed, visually interpreted, qualitative immunoassay based on Rapid Vertical Flow Technology® for the detection of antibodies to Treponema pallidum (TP), the causative agent of syphilis, and to nontreponemal (nTP; [RPR titer ≥ 1:8]) antigens in human serum, plasma, or fingerstick whole blood specimens. Nontreponemal antibodies are called reagins and they are generated after the tissue damage caused by syphilis infection.
  Multiplo® TP/nTP is intended for use by healthcare professionals as an aid in the diagnosis of active syphilis infection.
  Arms: Patients

SUMMARY:
The goal of this clinical trial is to implement a test, treat, and connect intervention approach using HIV and syphilis rapid point-of-care (POC) testing in 3 Canadian Prairie provinces (Alberta, Manitoba, and Saskatchewan), reaching 10,000 people in underserved communities.

DETAILED DESCRIPTION:
The goal of this clinical trial is to implement a test, treat, and connect intervention approach using HIV and syphilis rapid point-of-care (POC) testing in 3 Canadian Prairie provinces (Alberta, Manitoba, and Saskatchewan), reaching 10,000 people in underserved communities.

The study aims to recruit 10,000 people who are attending clinics for routine sexually transmitted and blood-borne testing in those provinces with opportunities for them to receive immediate treatment for syphilis, and culturally appropriate care and treatment for syphilis and HIV.

The primary objective is develop, implement and evaluate community-based models for "testing, treatment and linkages to care" for HIV and syphilis for those who are undiagnosed and underserved in the Prairie provinces.

The secondary objectives are:

Evaluate diagnostic performance of the investigational syphilis standalone POC test to standard testing.

Test the accuracy and usability of the investigational syphilis standalone POC test by intended users.

Assess the impact of POC testing on time to diagnosis, treatment, and connect to a clinical provider.

Investigate the feasibility and acceptability of the POC test among healthcare providers and at-risk populations.

Examine the acceptability of syphilis and HIV POC tests among at-risk and underserved populations.

Critical to the success of this, the study will engage and support people with lived experiences, peer navigators and leaders from community-based agencies to be involved in all aspects of this work.

ELIGIBILITY:
Test participants:

Inclusion Criteria:

1. Individuals > 16 years old accessing STBBI testing at specific locations
2. Able to provide informed consent.

Due to the number of sites across SK, AB, and MB, the diversity of the sites and local teams and the incremental addition of sites as the project progresses, the total number of participants to be recruited over the duration of the study (3 years), will be 10,000 individuals and there will be no requirement on local sample size, for the participating sites. (Please refer to Risks and Benefits). A competitive recruitment process will be in place and monitored closely throughout the study.

Exclusion Criteria:

1. < 16 years
2. Unable to provide signed informed consent (e.g., intoxicated)

Non-Healthcare Professional Operators For the purposes of this study, the untrained non-HCP operators are defined as the personnel, including community health navigators who in the opinion of the Principal Investigator are able to perform the study procedures outlined in this protocol and who are employed by the site. These operators will only be using the investigational device in this study - Multiplo® Complete Syphilis point-of-care test.

Inclusion criteria:

1. Individuals > 18 years old
2. Are able to read/understand English or French
3. Are able to provide informed consent
4. Are paid employees of the study site(s)
5. Are able to perform the study procedures outlined in the protocol

Exclusion criteria:

1. Individuals < 18 years old
2. Have used or watched someone use the Multiplo® Complete Syphilis Test prior to this study
3. Are regulated healthcare professionals including nurses, nurse practitioners, physicians, dentists, pharmacists, and laboratory technologists

Healthcare Professional Operators For the purposes of this study, the healthcare professionals are defined as the paid personnel who in the opinion of the Principal Investigator are able to perform the study procedures outlined in this protocol and who are employed by the site.

Inclusion criteria:

1. Regulated healthcare professional
2. Are able to read/understand English or French
3. Are able to provide informed consent
4. Are paid employees of the study site(s)
5. Are able to perform the study procedures outlined in the protocol

Exclusion criteria:

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of True Positives and True Negatives in Point-of-Care Syphilis Testing Compared to Standard Laboratory Testing (Sensitivity and Specificity Analysis) | 3 years
  Diagnostic performance of POC T Pallidum antibody and non-T Pallidum antibody test results will be compared to standard laboratory testing results for each marker, and test performance characteristics with 95% binomial confidence intervals will be calculated for sensitivity and specificity. In addition, diagnostic performance for TP antibody detection will be stratified by RPR titre (non-reactive, 1:1, 1:2, 1:4, >1:8 dilutions). Serial, parallel serology will be collected at the time of every syphilis POCT. Serology is the gold standard to diagnose syphilis and aids in determining staging and thus, treatment. Serial testing will aid whether syphilis POCT may be utilized in a more comprehensive manner, to possibly replace serology in some settings where access may be a challenge.

SECONDARY OUTCOMES:
Time to Diagnosis, Treatment, and Linkage to HIV Care Following Point-of-Care Testing vs. Standard Testing | 3 years
  Assess the time to diagnosis, time to treatment, and time to HIV care linkage following point-of-care testing for syphilis and HIV compared to standard laboratory testing. Time to diagnosis and treatment will be measured in days from test administration to diagnosis and from diagnosis to treatment, respectively. For HIV, time to linkage to care will be measured in days from diagnosis to first consultation with an infectious disease specialist.
  Data will be stratified by age, gender, and testing location, and analyzed using survival analysis or Poisson/negative binomial regression. Comparisons will be made between POC and standard testing with statistical significance determined by a p-value of <0.05.
Proportion of Patient Consenting vs. Declining (Patient Acceptability of Point-of-Care Testing ) | 3 years
  To evaluate the acceptability and feasibility of POC among different populations for syphilis (and HIV if applicable) among at risk and underserved populations, specifically patient acceptability and experiences with POC.
  Patient acceptability will be calculated as the proportion of individuals consenting to POCT divided by the total number of participants offered POC testing. To determine differences between participants consenting and those declining POC testing, age, gender, and testing location will be compared using chi-square for categorical variables and Mann-Whitney U test for age. A two-sided p value of < 0.05 will be considered statistically significant.
Descriptive Analysis of Healthcare Provider Feasibility and Acceptability of Point-of-Care Testing | 3 years
  Healthcare providers will complete a survey after point-of-care testing assessing their experience using the test (e.g., ease of use, ease of interpretation of results). A descriptive analysis of healthcare provider experience survey will be conducted.
Descriptive Analysis of Patient Experience and Satisfaction of Point-of-Care Testing | 3 years
  Patients will complete a survey after point-of-care testing assessing their experience (e.g., comfort levels, recommend to others, ease of testing process).
  A descriptive analysis of the patient experience survey will be completed and stratified by negative and positive results by test type.
Demographic Associations with Syphilis and HIV Point-of-Care Test Outcomes (Reactive vs. Non-Reactive Results) | 3 years
  Analyze the associations between demographic factors (such as age, gender, and testing location) and syphilis and HIV point-of-care test outcomes, focusing on the correlation between demographics and reactive versus non-reactive test results. Chi-square analysis will be used to assess these associations, with stratification by POC test type when sample sizes allow. A two-sided p-value of <0.05 will be considered statistically significant.

CONTACTS AND LOCATIONS:
Locations (8):
- Canada (8):
  - Radius Community Health & Healing, Edmonton, Alberta
  - StreetWorks, Edmonton, Alberta
  - Northreach Society, Grande Prairie, Alberta
  - Siloam Mission, Winnipeg, Manitoba
  - Ka Ni Kanichihk, Winnipeg, Manitoba
  - Nine Circles Community Health Centre, Winnipeg, Manitoba
  - All Nations Hope Network, Regina, Saskatchewan
  - Wellness Wheel Clinic, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No